CLINICAL TRIAL: NCT06834425
Title: Efficacy of NSAID Peritendinous Injection for Acute Tendinitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Yu-Hsuan Cheng, Department of Physical Medicine and Rehabilitation, Wan-Fang Hospital, Taipei Medical Univerisity, Taipei Medical University WanFang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N202412008; 114-wf-eva-19 (Other Grant/Funding Number: Wan Fang Hospital, Taipei Medical University)
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Tendinitis; Acute Tendonitis; NSAID (Non-Steroidal Anti-Inflammatory Drug)
MeSH Terms: conditions — Tendinopathy | interventions — Anti-Inflammatory Agents, Non-Steroidal; Control Groups; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Local anesthetics and NSAID(parecoxib) peritendinous Injection for acute tendinitis
  Interventions: Drug: Peritendinous NSAID injection
- Control group (Placebo Comparator): Local anesthetics and normal saline peritendinous injection for acute tendinitis
  Interventions: Drug: Control group (placebo)

INTERVENTIONS:
Drug: Peritendinous NSAID injection — Peritendinous NSAID (parecoxib) injection
  Other Names: NSAID injection
  Arms: Intervention group
Drug: Control group (placebo) — Normal saline mixed with local anesthetics injection
  Other Names: Sham injection
  Arms: Control group

SUMMARY:
This study evaluates whether NSAID peritendinous or ligament injections at acute sprain sites can relieve pain and restore function.

Forty patients will be randomly assigned to either the injection or oral NSAID group. Pain will be assessed subjectively using the Numeric Pain Rating Scale and objectively through pressure pain threshold measurements. Functional outcomes (DASH for the upper limb, FADI for the lower limb) will be evaluated before treatment and at 3 days, 1 week, and 4 weeks post-treatment.

DETAILED DESCRIPTION:
Acute tendon inflammation is a common sports injury, typically treated with oral or topical non-steroidal anti-inflammatory drugs (NSAIDs) or local corticosteroid injections at the affected site. Direct corticosteroid injections provide the fastest relief; however, the World Anti-Doping Agency (WADA) has restricted the use of corticosteroids by any route in its latest banned substance list. As a result, corticosteroid injections into tendons or joints, which were previously allowed during competitions, can no longer be used. Currently, the only methods available for acute inflammation relief during competitions are oral NSAIDs and ice therapy. For athletes without structural damage who need to quickly reduce inflammation and return to play, these methods may be insufficient.

Previous clinical studies on NSAID injections into tendons and joints have shown that local NSAID injections are equally effective as corticosteroid injections for treating shoulder impingement syndrome and knee osteoarthritis. However, these studies mainly focused on patients with chronic arthritis and tendinitis. The difference in efficacy between oral NSAIDs and tendon injections during the acute phase of inflammation remains unknown. This study aims to compare different routes of NSAID administration to identify the most appropriate treatment for managing acute tendinitis in high-level athletes.

We hypothesize that peritendinous NSAID injections will provide greater pain relief and functional improvement.

ELIGIBILITY:
Inclusion Criteria:

* Ultrasonography diagnosed acute tendinitis with inflammation
* 20-70 years old

Exclusion Criteria:

* Cognitive impairment.
* Post operation at painful site.
* Neuropathic pain or vascularity disease
* Unable to receive injection therapy, including a history of syncope during injection.
* Allergy history to NSAID
* Within 14 days after coronary artery bypass graft, CABG

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | Baseline, at 12 hours post-injection, and on each day from 1 to 7 days after the injection.
  The 11-point Numeric Rating Scale (NRS) is a subjective pain assessment tool that ranges from 0 to 10. A score of '0' indicates the complete absence of pain (e.g., "no pain"), while a score of '10' represents the most severe pain imaginable (e.g., "pain as bad as you can imagine" or "worst pain imaginable"). This scale allows individuals to quantify their pain intensity, facilitating communication between patients and healthcare providers for better pain management.

SECONDARY OUTCOMES:
Disabilities of the Arm, Shoulder, and Hand (DASH) | Baseline, 3-day, 7-day and 28-day after injection
  Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire for upper limb functionality
Foot and Ankle Disability Index (FADI) | Baseline, 3-day, 7-day and 28-day after injection
  Foot and Ankle Disability Index (FADI) for lower limb functionality.
Pain pressure threshold | Baseline, 3-day, 7-day and 28-day after injection
  A manometer was used to measure the pain pressure threshold at the most tender point of the affected area.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsuan Cheng, MD, MS, Study Chair — Taipei Medical University
Locations (1):
- Wan Fang Hospital, Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rhim HC, Ruiz J, Taseh A, Afunugo W, Crockett Z, Schon J, Pan X, Shin J, Schowalter S, Jang KM, Robinson DM. Nonsteroidal Anti-Inflammatory Drug Injections versus Steroid Injections in the Management of Upper and Lower Extremity Orthopedic Conditions: A Systematic Review with Meta-Analysis. J Clin Med. 2024 Feb 17;13(4):1132. doi: 10.3390/jcm13041132. PMID 38398445
- [Result] Ziradkar R, Best TM, Quintero D, Paultre K. Nonsteroidal Anti-inflammatory and Corticosteroid Injections for Shoulder Impingement Syndrome: A Systematic Review and Meta-analysis. Sports Health. 2023 Jul-Aug;15(4):579-591. doi: 10.1177/19417381221108726. Epub 2022 Jul 27. PMID 35897160
- [Result] Sardana V, Burzynski J, Hasan K, Zalzal P. Are non-steroidal anti-inflammatory drug injections an alternative to steroid injections for musculoskeletal pain?: A systematic review. J Orthop. 2018 Aug 16;15(3):812-816. doi: 10.1016/j.jor.2018.08.022. eCollection 2018 Sep. PMID 30140124
- [Result] Kim YB, Lee WS, Won JS. The effects of a single-dose subacromial injection of a nonsteroidal anti-inflammatory drug in geriatric patients with subacromial impingement syndrome: a randomized double-blind study. Clin Shoulder Elb. 2021 Mar;24(1):4-8. doi: 10.5397/cise.2021.00052. Epub 2021 Mar 2. PMID 33652505
- [Result] Bellamy JL, Goff BJ, Sayeed SA. Economic Impact of Ketorolac vs Corticosteroid Intra-Articular Knee Injections for Osteoarthritis: A Randomized, Double-Blind, Prospective Study. J Arthroplasty. 2016 Sep;31(9 Suppl):293-7. doi: 10.1016/j.arth.2016.05.015. Epub 2016 May 18. PMID 27402605
- [Result] Min KS, St Pierre P, Ryan PM, Marchant BG, Wilson CJ, Arrington ED. A double-blind randomized controlled trial comparing the effects of subacromial injection with corticosteroid versus NSAID in patients with shoulder impingement syndrome. J Shoulder Elbow Surg. 2013 May;22(5):595-601. doi: 10.1016/j.jse.2012.08.026. Epub 2012 Nov 22. PMID 23177167
- [Result] Shakeel H, Ahmad TS. Steroid injection versus NSAID injection for trigger finger: a comparative study of early outcomes. J Hand Surg Am. 2012 Jul;37(7):1319-23. doi: 10.1016/j.jhsa.2012.03.040. PMID 22721455